CLINICAL TRIAL: NCT06207201
Title: Discover In-Hospital Cardiac Arrest: A Prospective Multicenter Study of Post-In-Hospital Cardiac Arrest Management Practices
Brief Title: Discover In-Hospital Cardiac Arrest
Acronym: Discover IHCA
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Society of Critical Care Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-14602
Record Dates: First submitted 2023-12-20; First posted 2024-01-16 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Arrest
Keywords: In-hospital cardiac arrest; Post-cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Discover In-Hospital Cardiac Arrest (IHCA) study is a multicenter, prospective observational study aimed at better understanding variations in practice for the post-in-hospital cardiac arrest patient.

DETAILED DESCRIPTION:
There is considerable debate among experts concerning many components of intra- and post-arrest care. This study aims to increase the evidence base of these components, particularly temperature control, and prognostication in post-in-hospital cardiac arrest patients. In addition to providing insights regarding immediate and long-term post-arrest care, data collected will also be useful in studying variations in cardiopulmonary resuscitation practices.

This project is endorsed by the Society of Critical Care Medicine's (SCCM) Discovery, the Critical Care Research Network.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old) patients
* Patients with a cardiac arrest (a lack of palpable pulse or perfusing cardiac activity) while admitted to the hospital
* Patients admitted to a ward (telemetry or non-telemetry) or an intensive care unit, or are admitted but still in the emergency department waiting for a hospital bed
* Patients who achieved return of spontaneous circulation (ROSC defined as >20 minutes of sustained spontaneous circulation) OR initiated on extracorporeal membrane oxygenation (eCPR) with chest compressions ongoing
* Patients survived for 6 hours after ROSC

Exclusion Criteria:

* Cardiac arrest in non-inpatients (e.g. outpatients, visitors)
* Patients whose cardiopulmonary resuscitation (CPR) starts outside of the hospital
* Non-index arrests (arrests that are not the patient's first arrest during the hospital admission; this also excludes patients who were initially admitted for an out-of-hospital cardiac arrest)
* Patients suffering IHCA in the operating room (OR) or post anesthesia care unit (PACU)
* Patients with cardiac arrest after arriving to an emergency department (ED) but prior to being evaluated and admitted to the hospital
* Cardiac arrests lasting <2 minutes (i.e. chest compressions performed <2 minutes)
* Cardiac arrests where the patient is transitioned to comfort focused care within 6 hours of return of spontaneous circulation (ROSC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult index in-hospital cardiac arrests where ROSC is achieved for > 6 hours and the patient is not transitioned to comfort care in the first 6 hours after ROSC.
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Fever Incidence | Up to 96-hours post cardiac arrest
  The incidence of fever from ROSC until 96 hours after ROSC among patients who remain comatose
Multimodal Prognostication | Up to 60 days post cardiac arrest
  The use of at least two approaches for prognostication prior to withdrawal of care from ROSC until hospital discharge
Early Withdrawal of Care | Up to 72-hours post cardiac arrest
  The withdrawal of care from ROSC until 72-hour after ROSC

CONTACTS AND LOCATIONS:
Overall Officials: Ari Moskowitz, MD, MPH, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No